CLINICAL TRIAL: NCT04049435
Title: Assessment of Horizontal Bone Gain Using Patient Specific Titanium Sheet: a Novel Protocol for Treatment of Horizontal Deficiency in the Anterior Maxilla (Case Series Study ).
Brief Title: Horizontal Bone Gain Using Titanium Sheet (Case Series Study ).
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdelwakeel mohamed abdelrahman hamam, Assessment of Horizontal Bone gain using patient specific titanium sheet: a novel protocol for treatment of horizontal deficiency in the anterior maxilla (Case series study )., Cairo University
Other Study IDs: OMFS 3-3-14
Record Dates: First submitted 2019-08-02; First posted 2019-08-08 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Anterior Teeth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- horizontal deficiency anterior maxilla: Using the titanium sheet in augmentation of horizontally deficient anterior maxilla will be efficient, time saving, accurate reconstruction
  Interventions: Device: Assessment of Horizontal Bone gain using patient specific titanium sheet: a novel protocol for treatment of horizontal deficiency in the anterior maxilla

INTERVENTIONS:
Device: Assessment of Horizontal Bone gain using patient specific titanium sheet: a novel protocol for treatment of horizontal deficiency in the anterior maxilla — Assessment of Horizontal Bone gain using patient specific titanium sheet: a novel protocol for treatment of horizontal deficiency in the anterior maxilla

SUMMARY:
The horizontal deficient anterior maxilla less than 3mm presents considerable challenges for surgical and prosthetic reconstruction. caused by trauma , infection, congenitally missing teeth or resorption subsequent to dental extractions hampers dental implant placement(Aghaloo & Moy, 2007)

DETAILED DESCRIPTION:
The successful use of dental implants for replacing missing dentition requires adequate available bone in the treatment planning phase and inserting the implant in the correct 3D position to achieve good esthetic and function outcomes.(Rieder et al., 2016)

The horizontal deficient anterior maxilla presents considerable challenges for surgical and prosthetic reconstruction. Inadequate alveolar ridge width caused by trauma , infection, congenitally missing teeth or resorption subsequent to dental extractions hampers dental implant placement (Aghaloo & Moy, 2007)

Avariety of bone augmentation technigue have been described to enhance the bone volume of the deficient implant recipient site such as autogenous bone graft ,synthetic bone graft ,distraction osteogenesis ,ridge splitting, guided bone regeneration(Rakhmatia, Ayukawa, Furuhashi, & Koyano, 2013)(Gulinelli et al., 2017)

Autograft remain the gold standard with the capacity to regenerate and forming new bone through its osteogenic ,osteoconductive and osteoinductive properties which can be obtained from chin area (Donos, Mardas, & Chadha, 2008).

Due to the limited availabity of autograft in case of sever resorped ridge ,xenogrft can be mixed to increase the amount of bone applied to the defective area(Monje et al., 2015)

However considerable graft resorption following augmentation and the graft was not sufficiently stable during the healing period ,the titanium membrane or sheet used to overcome this problem(Andreasi Bassi et al., 2016)

The titanium sheet is non resorbable membrane , impermeable ,rigid acts as space maintainance, clot protection , a barrier preventing bacterial contamination of the gaft , stopping the graft resorption , less morbid,less operative time , more accurate for contour reconstruction than the well known autogenous bone technique (Andreasi Bassi et al., 2016)

Computer aided design/computer aided manufacturing technology (CAD/CAM) have been established in creation of three dimensional(3D) framework , Digitally virtually planned regenerated ridge was created from a cone-beam computerized tomography (CBCT) using specialized DICOM image ( Digital imaging and communication in medicine reconstructing 3D surgical model, and the design of the titanium sheet with the location of the bone screws was preserved. The new 3D surgical model with the simulated surgery was used to fabricate titanium sheet positioning with all required dimensions decreasing the overall operative time .(Al-Ardah et al., 2018)

The quality of newly formed bone will be evaluated by histologically at the time of implant placement , core biopsies will be retrieved . the specimen will immediately fixed in 10% buffered formalin for 1 week, then decalcified and processed according to standardized protocol Ethylenediamine-tetracetic acid (EDTA)-formic acid combination differentiating the newly formed bone end from the native bone end for histologic analysis(Atef, Hakam, Elfaramawey, Abou-Elfetouh, & Ekram, 2014)

Following postoperative healing period of 6 months CBCT scan will take to evaluate the horizontal bone gain and planning of implant surgery(Mendoza-Azpur, Fuente, Chavez, Valdivia, & Khouly, 2019)

ELIGIBILITY:
Inclusion Criteria:

1. Horizontal deficient anterior maxilla < 3mm.
2. All ages >18 years

Exclusion Criteria:

- 1. Patients systemic disease or immunocomprmized status that may affect normal healing of bone, and predictable outcome.

2. Patients with history of previous grafting procedure 3. Patients with physical and psychological intolerance

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Case series
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2019-09-25 (Estimated); Primary Completion 2020-10-31 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Horizontal bone gain | after 6 months
  Distanc buccolingually

SECONDARY OUTCOMES:
Gained bone quality measured by histomorphomerty examination of core biopsy | after 6 months
  Histomorphometry of core biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Abdelwakeel Mohammed, Principal Investigator — Investigator
Locations (1):
- Abdelwakeel, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Undecided: It is not yet known if there will be a plan to make IPD available.
Supporting Information: Study Protocol
Time Frame: 2years
Access Criteria: This study will carried out on patients attending clinic of Master program for Oral Implantology - Faculty of Dentistry Cairo University.

REFERENCES:
- [Result] Aghaloo TL, Moy PK. Which hard tissue augmentation techniques are the most successful in furnishing bony support for implant placement? Int J Oral Maxillofac Implants. 2007;22 Suppl:49-70. PMID 18437791